CLINICAL TRIAL: NCT00337987
Title: A Pilot Phase II Study to Determine the Safety of the Combination of ONTAK (DAB389IL-2), an Interleukin-2 Fusion Toxin, in Combination With CHOP in Peripheral T-Cell Lymphoma
Brief Title: A Pilot Study to Determine the Safety of the Combination of Ontak in Combination With CHOP in Peripheral T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0507000369
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — denileukin diftitox; Cyclophosphamide; Doxorubicin; Protons; Vincristine; Prednisone; Drug Therapy

INTERVENTIONS:
Drug: Ontak — ONTAK ( denileukin diftitox) is given at 18 mcg/kg/d (Days 1,2) plus CHOP therapy (Day 3) q 21 days x 6 cycles (cyclophosphamide 750 mg/m²IV, doxorubicin 50 mg/m²IV day, vincristine 1.4 mg/m²IV day, and prednisone 100 mg q day PO days #3-7) plus, G-CSF support beginning on Day 4 to prevent neutropenia
  Other Names: DAB 389 IL-2
Drug: CHOP (cyclophosphamide (C), adriamycin (H), vincristine (O), and prednisone (P)) chemotherapy — ONTAK ( denileukin diftitox) is given at 18 mcg/kg/d (Days 1,2) plus CHOP therapy (Day 3) q 21 days x 6 cycles (cyclophosphamide 750 mg/m²IV, doxorubicin 50 mg/m²IV day, vincristine 1.4 mg/m²IV day, and prednisone 100 mg q day PO days #3-7) plus, G-CSF support beginning on Day 4 to prevent neutropenia

SUMMARY:
The standard treatment for PTCL is CHOP (cyclophosphamide (C), adriamycin (H), vincristine (O), and prednisone (P)) chemotherapy. This study is attempting to determine whether adding other treatments to CHOP therapy will improve the chance of the disease going into remission or staying in remission. Because other drugs for T-cell lymphoma have not yet been given with CHOP, this study is looking at combining CHOP with ONTAK. ONTAK has been FDA approved for treatment of Cutaneous T cell Lymphoma and works by specifically binding to a protein on the surface of the tumor cells and killing the cell without causing damage to other types of cells in the body. Studies have shown that ONTAK has helped patients with PTCL who have failed chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of peripheral T-cell lymphoma of one of following histologies as per the REAL classification: peripheral T-cell lymphoma (unspecified), anaplastic large cell lymphoma CD30+, angioimmunoblastic T-cell lymphoma, nasal/nasal type T/NK cell lymphoma, intestinal T-cell lymphoma, hepatosplenic T-cell lymphoma, subcutaneous panniculitic T-cell lymphoma.
* Treatment naive except for prior radiation or a single cycle of CHOP.
* Patients must have at least one clear-cut bidimensionally measurable site by physical exam and/or computed tomography. Baseline measurements of measurable sites and evaluation of evaluable disease must be obtained within 4 weeks prior to registration to this study.
* Prior radiation therapy for localized disease is allowed as long as the irradiated area is not at the mediastinal area or at the only site of measurable disease. Therapy must be completed at least 4 weeks before the enrollment in study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Age > 18 years old.
* Adequate bone marrow reserve, indicated by absolute neutrophil count (ANC) ≥ 1000/mm³, platelets ≥50,000/mm³(25,000/mm³ if thrombocytopenia secondary to bone marrow involvement by lymphoma), and hemoglobin ≥8 g/dL. These values must be obtained within 2 weeks before protocol entry.
* Adequate liver function, indicated by bilirubin ≤1.5 times the upper limit of normal (ULN), alanine transaminase (ALT) ≤2 times the ULN or aspartate transaminase (AST) ≤2.0 times the ULN and albumin > 3.0 g/dl.
* Adequate renal function, indicated by serum creatinine ≤2.5 mg/dL. Laboratory values must be obtained within 2 weeks before study entry.
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception.
* Able to give informed consent.

Exclusion Criteria:

* Patients with diagnosis of Mycosis Fungoides or Sezary Syndrome
* Patients with active Hepatitis B or Hepatitis C infection.
* Patients with known HIV infection are excluded. These patients are excluded because the potential to target activated T-cells, in a population of patients already at risk for T-cell depletion, would be a contraindication to therapy. HIV testing is not required.
* Patients with active infections requiring specific anti-infective therapy are not eligible until all signs of infections are resolved and any continuing treatment is given on an outpatient basis.
* Patients with previous anthracycline therapy (cumulative dose of > 100 mg/m2).
* Patients with Left Ventricular Ejection Fraction (LVEF) < 50%.
* Patients who are pregnant or breast-feeding. These patients are excluded because the effects of this treatment on the fetus and young children are unknown.
* Prior invasive malignancies within past 5 years.
* Allergic to or history of allergy to diphtheria toxin or IL-2.
* Preexisting severe cardiovascular disease (e.g. CHF, Severe CAD, cardiomyopathy, MI within past 3 months, arrhythmia) requiring ongoing treatment.
* Ongoing antineoplastic chemotherapy, radiation, hormonal (excluding contraceptives) or immunotherapy, or investigational medications within past 30 days.
* Patients with deep vein thrombosis within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francine Foss, M.D., Principal Investigator — Yale University
Locations (1):
- Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Denileukin Diftitox/CHOP Administration: Patients received six 21-day cycles of therapy, up to a maximum of 8 cycle. Each cycle comprised of denileukin diftitox plus CHOP (cyclophasphamide, doxorubicin, vincristine, prednisone)
Period: Overall Study
Arm/Group | Denileukin Diftitox/CHOP Administration
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Denileukin Diftitox/CHOP Administration
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 52 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Achieved a Complete Response or a Partial Response (PR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: After 4 years
Measure: Number; unit: participants
Arm/Group | Denileukin Diftitox/CHOP Administration
Number analyzed (Participants) | 49
participants | 32

2. Primary Outcome: Number of Patients That Achieved a Complete Response (CR)
Description: as for outcome 1
Time Frame: After 4 years
Measure: Number; unit: participants
Arm/Group | Denileukin Diftitox/CHOP Administration
Number analyzed (Participants) | 49
participants | 27

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Denileukin Diftitox/CHOP Administration
Serious Adverse Events (participants affected / at risk) | 25/49
Other Adverse Events (participants affected / at risk) | 42/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denileukin Diftitox/CHOP Administration (N=49)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5
Fever (General disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 4
Allergic Reaction/Allergy (Immune system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Cardiac Arrest (Cardiac disorders) | 3
Death NOS (General disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denileukin Diftitox/CHOP Administration (N=49)
Anemia (Blood and lymphatic system disorders) | 20
Leukocytopenia (Blood and lymphatic system disorders) | 17
Lymphopenia (Blood and lymphatic system disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 13
Fatigue (General disorders) | 31
Nausea (Gastrointestinal disorders) | 23
Neuropathy, sensory (Musculoskeletal and connective tissue disorders) | 20
Alanine Aminotransferase (ALT) Elevated (Blood and lymphatic system disorders) | 17
Hyperglycemia (Metabolism and nutrition disorders) | 17
Hypoalbuminemia (Hepatobiliary disorders) | 17
Fever (General disorders) | 16
Hypocalcemia (Metabolism and nutrition disorders) | 15
Aspartate Aminotransferase (AST) Elevation (Hepatobiliary disorders) | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14
Alopecia (Skin and subcutaneous tissue disorders) | 13
Constipation (Gastrointestinal disorders) | 12
Edema, peripheral (Vascular disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 10
Dysgeusia (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Heartburn (Gastrointestinal disorders) | 8
Bone Pain (General disorders) | 8
Vomiting (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes